CLINICAL TRIAL: NCT03229018
Title: Effect of Different Voxel Sizes on Accuracy of 2D and 3D Mandibular Linear Measurements Using CRANEX® 3D Cone Beam Computed Tomography Machine: Preclinical Study
Brief Title: Effect of Different Voxel Sizes on Accuracy of CBCT Linear Measurements: Preclinical Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Mohamed Selim, Master student, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1611
Record Dates: First submitted 2017-07-13; First posted 2017-07-25 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Cone-Beam Computed Tomography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- voxel size (Other): 200 μm and 300 μm Voxel Sizes
  Interventions: Diagnostic Test: Voxel size

INTERVENTIONS:
Diagnostic Test: Voxel size — 200 μm and 300 μm Voxel Sizes

SUMMARY:
study target is assessment of the accuracy of linear measurement obtained from CBCT images on 3D volumetric rendering and multiplanar slices with different voxel sizes

DETAILED DESCRIPTION:
The real linear measurement will be measured in millimeter (mm) on the mandibles using digital caliper in the chosen areas.

CBCT images will be viewed by OnDemand3D™ viewer software and linear measurements using 2D ruler on multiplanar slices and 3D ruler on 3D volumetric rendering to assess for the dimension in the chosen areas.

ELIGIBILITY:
Inclusion Criteria:

* Selection of the human dry mandibles will be independent of age, gender and ethnicity.
* They should be intact, free from any bone defects, fractures, pathology.
* Dentate state of the mandibles is not an element in selection criteria; either dentulous or edentulous mandibles are acceptable

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of linear measurement | 1 year
  Assessment of the accuracy of linear measurement obtained from CBCT images on 3D volumetric rendering and multiplanar slices with different voxel sizes

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No